CLINICAL TRIAL: NCT02175797
Title: Assessment of the MRI Solution: KORA 100 and Beflex Pacing Leads System
Acronym: IKONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MicroPort CRM (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IBMR02 - IKONE
Record Dates: First submitted 2014-06-04; First posted 2014-06-26 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Bradycardia
Keywords: Pacemaker, leads and MRI exam
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pacemaker + leads (Other): all patients must have a MRI exam after pacemaker implantation
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — at least 6 weeks after the implantation of the pacemaker a MRI exam is performed

SUMMARY:
The purpose of this study is to report the stability of atrial and ventricular leads by absence of effect of the MRI exam on the pacing and sensing threshold and to report the safety based on the serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patient who is already implanted with following system KORA 100 (SR or DR) pacemaker and Beflex RF45D and/or RF46D pacing leads in the left or right pectoral region
* Patient who is able and willing out-of-chest non medical indicated MRI scanning OR patients with planned medical indicated out of chest MRI scanning
* Patient who fulfils MRI solutions conditions
* Patient who provides signed and dated informed consent

Exclusion Criteria:

* Implanted or planned to be implanted non MR-compatible device or material
* Permanent Atrial Fibrillation (for DR devices)
* Diaphragmatic/phrenic stimulation
* Claustrophobia
* Incessant ventricular tachyarrhythmia
* Inability to understand the purpose of the study or refusal to co-operate
* Unavailability for scheduled follow-ups at the implanting centre
* Already included in another clinical trial that could affect the results of this study
* Patient is minor (less than 18-years old)
* Patient is pregnant - Patient is forfeiture of freedom or under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Measure the atrial and ventricular pacing thresholds in Volts before and after the MRI exam, using the programmer. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Mr SAVOURE, cardiologist, Principal Investigator — CHU Charles Nicolle - 1 rue Germont, 76000 ROUEN
Locations (1):
- CHU Charles Nicolle, Rouen, France